CLINICAL TRIAL: NCT06848907
Title: Re Evaluation of the Clinical Efficacy of Ganzhixiao Capsules Based on MRI-PDFF in the Treatment of Metabolic Related Fatty Liver Disease
Brief Title: Clinical Study on the Treatment of MAFLD With Ganzhixiao Capsules
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dong Hui (Other)
Responsible Party: Sponsor-Investigator, Dong Hui, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TJ-IRB202504027
Record Dates: First submitted 2025-02-15; First posted 2025-02-27 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: MAFLD

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinical study on the treatment of MAFLD with palcebo capsules (Placebo Comparator)
  Interventions: Drug: placebo capsule
- Clinical study on the treatment of MAFLD with Ganzhixiao capsules (Experimental)
  Interventions: Drug: ganzhixiao capsule

INTERVENTIONS:
Drug: ganzhixiao capsule — Ganzhixiao Capsule is mainly composed of Bupleurum chinense, Herba Artemisiae, Polygonum cuspidatum, Rhubarb and Hawthorn.Take 3 capsules each in the morning, afternoon, and evening, and swallow with warm water after meals for 16 weeks.All participants in the trial were required to have a low-fat diet and engage in aerobic exercise for 150 minutes per week.
  Arms: Clinical study on the treatment of MAFLD with Ganzhixiao capsules
Drug: placebo capsule — Take 3 palcebo capsule each in the morning, afternoon, and evening, and swallow with warm water after meals for 16 weeks.All participants in the trial were required to have a low-fat diet and engage in aerobic exercise for 150 minutes per week.
  Arms: Clinical study on the treatment of MAFLD with palcebo capsules

SUMMARY:
This trial is expected to enroll 138 MAFLD patients in one clinical center, who will be randomly divided into a placebo group and a Ganzhixiao capsule group in a 1:1 ratio. There will be 69 patients in the Ganzhixiao group and 69 patients in the placebo group. Administer Ganzhixiao capsules or mimetics separately, intervene for 16 weeks, and compare the liver fat content、 ALT、 Changes in indicators such as cytokeratin 18 fragment, FIB-4 score, and LSM score. Among them, MRI-PDFF is the main efficacy evaluation index to evaluate the clinical efficacy of Ganzhixiao capsules in the treatment of MAFLD.

DETAILED DESCRIPTION:
All participants in the trial were required to have a low-fat diet and engage in aerobic exercise for 150 minutes per week.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years old, with a body mass index (BMI) of at least 24kg/m2;
* Diagnosis of NAFLD determined by imaging [ultrasound, computed tomography or magnetic resonance imaging (MRI-PDFF)] or liver biopsy, showing MAFLD or simple steatosis within the last 24 months prior to screening;
* MAFLD patients conform to the damp heat syndrome type; ④ Voluntary signing of informed consent form

Exclusion Criteria:

* Blood biochemical indicators ALT, AST, BUN are greater than 1.5 times the upper limit of normal values, Cr is greater than the upper limit of normal values, eGFR<60ml/min/1.73m2;
* Alcoholic fatty liver, other chronic liver diseases, cirrhosis, liver malignant tumors, etc.;
* Type 2 diabetes and pancreatic diseases;
* Taking some hypoglycemic, lipid-lowering, liver protective drugs or high-dose vitamin E that may affect the efficacy judgment in the past three months;
* Patients with severe infections, cardiovascular, respiratory, renal, hematological, rheumatic connective tissue disease, neuropsychiatric, and non liver malignant tumors;
* Pregnant or lactating women;
* Those who require long-term hormone therapy;
* Researchers anticipate poor compliance or inability to cooperate;
* There are contraindications for MRI examination, including pacemakers or cochlear implants, postoperative artificial valve replacement, presence of ferromagnetic vascular clips in the body, metal foreign bodies in the eyeball, insulin pumps, ferromagnetic objects in the scanning field, metal dentures, intrauterine devices, and patients with claustrophobia.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2025-05-30 (Estimated); Primary Completion 2028-05-30 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
MRI-PDFF | 16 weeks
  MRI PDFF (Magnetic Resonance Proton Density Fat Fraction) is a non-invasive magnetic resonance technique used to evaluate the fat content of the liver. It reflects the concentration of free TG in tissues by measuring the ratio of the proton density of free TG to the total proton density of free TG and water, expressed as a percentage (%).

SECONDARY OUTCOMES:
ALT | 16 weeks
  ALT (Alanine Aminotransferase) is an indicator that can reflect liver function damage，which is measured in blood .
CK18 | 16 weeks
  Cell corner fragment 18 (CK18) is mainly used as a specific indicator for evaluating liver cell apoptosis, which can help us understand the degree and nature of liver damage. CK18 is measured in blood.
FIB-4 | 16 weeks
  The Fibrosis 4 Score (FIB-4) is a non-invasive indicator for assessing the degree of liver fibrosis in patients with chronic liver disease. This scoring system calculates the degree of liver fibrosis using simple blood indicators, including age, aspartate aminotransferase (AST), alanine aminotransferase (ALT), and platelet count (PLT).
LSM | 16 weeks
  The LSM score, also known as Liver Stiffness Measurement, is an indicator used to evaluate the degree of liver fibrosis through FibroScan.
body weight | 16 weeks
  body weight
waist circumference | 16 weeks
  waist circumference
hip circumference | 16 weeks
  hip circumference
waist to hip ratio | 16 weeks
  waist to hip ratio
Waist hip height ratio | 16 weeks
  Waist hip height ratio
Self-Rating Anxiety Scale | 16 weeks
  The Self Rating Anxiety Scale is used to assess an individual's anxiety symptoms
Self-rating depression scale | 16 weeks
  Self rating depression scale is used to assess an individual's depressive symptoms
Pittsburgh sleep quality index | 16 weeks
  Pittsburgh sleep quality index is used to evaluate an individual's sleep status
Damp Heat Traditional Chinese Medicine Syndrome Scale | 16 weeks
  Damp Heat Traditional Chinese Medicine Syndrome Scale is used to evaluate individual damp heat syndrome

IPD SHARING:
Plan to Share IPD: No